CLINICAL TRIAL: NCT01817439
Title: The Effect of Intravenous vs. Oral Administration of Amiodarone on the Incidence Rate of Phlebitis Among Patients With Recent Onset of Atrial Fibrillation (AF)
Brief Title: Safety and Efficacy of Oral Versus Intravenous Amiodarone in the Treatment of AF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, lilach shema, Coordinator, Quality Assurance Unit, Western Galilee Hospital-Nahariya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP 1
Record Dates: First submitted 2013-03-18; First posted 2013-03-25 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Atrial Fibrillation
Keywords: oral Amiodarone; IV Amiodarone; phlebitis; thrombophlebitis; adverse events
MeSH Terms: conditions — Atrial Fibrillation; Phlebitis; Thrombophlebitis | interventions — Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral amiodarone, group A (Experimental): oral amiodarone 400 mg three times a day for 2 days
  Interventions: Drug: Amiodarone
- IV amiodarone, Group B (Experimental): Amiodarone:
  IV loading of 300 mg for 30 min in 100cc glucose 5% IV infusion with 900 mg/24h in 1000cc glucose 5%
  Interventions: Drug: Amiodarone

INTERVENTIONS:
Drug: Amiodarone — patients will be randomly assigned to oral OR IV Amiodarone
  Other Names: Procor

SUMMARY:
Atrial fibrillation (AF) remains a significant contributor to cardiovascular morbidity. Amiodarone is a potent antiarrhythmic drug; however, patients receiving IV amiodarone are at high risk for phlebitis. Phlebitis may lead to infection, additional medical intervention, delay in treatment, and prolonged hospitalization. Therefore, examining new therapy approach, aimed to reduce the incidence of phlebitis is a valuable clinical and research goal.

Aim: To evaluate the safety and efficacy of oral versus intravenous (IV) Amiodarone in the treatment of AF of recent onset (duration < 48 h).

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common heart rhythm abnormality worldwide. Three therapeutic goals should be considered for each patient: Rate control, maintenance of sinus rhythm and prevention of thromboembolism. In managing AF, numerous antiarrhythmic drugs have been used. Intravenous amiodarone is a class III antiarrhythmic agent which has been reported to be safe and most effective in various clinical settings, without an associated increase in mortality rate. In most of the cases, the method of administration is via peripheral infusion. Phlebitis is the most common complication with peripheral infusion of amiodarone. Phlebitis adversely affects patient care; it may interfere with the continued infusion of amiodarone, necessitate insertion of another peripheral intravenous or central catheter, and extend hospitalization. Furthermore, patients who develop phlebitis, experience pain, swelling, and inflammation. Phlebitis can be prevented by oral administration.

The goal of the proposed study is to evaluate the incidence rate of phlebitis following IV administration of amiodarone and to investigate whether the oral administration of amiodarone in patients with recent onset AF (duration < 48 h), is safer than, and as efficient as, the IV administration of the same drug in the ICCU and ICU setting.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age,
* Patients who will be admitted to the ICCU / ICU wards
* Patients with recent onset of atrial fibrillation (duration < 48h).

Exclusion Criteria:

* Age < 18 years
* Baseline systolic blood pressure < 100 mm/hg
* Known thyroid disease
* Serum potassium < 3.5 mmol/l
* Pretreatment with amiodarone
* Pregnant or lactating women.
* Participation in other clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of phlebitis | during 24 h
  For detection of eventual amiodarone induced phlebitis the site of venous access will be examined 30 min, 3, 6, 12, 24 h after drug administration by one of the investigators

SECONDARY OUTCOMES:
incidence of hypotension | during 24 h
  blood pressure measurements will be taken on admission and during treatment at defined intervals of 3, 6, 12, 18 and 24 h
Cumulative incidence of restored sinus rhythm | During 48h
  Patients will be monitored during all stuffy period

CONTACTS AND LOCATIONS:
Overall Officials: Atar Shaul, MD, Principal Investigator — Western Galilee Hospital; Nicola Makhoul, MD, Principal Investigator — Western Galilee Hospital; Lilach Shema-didi, PhD, Principal Investigator — Western Galilee Hospital
Locations (1):
- Western Galilee Hospital, Nahariya, Israel, Israel